CLINICAL TRIAL: NCT07125599
Title: The Association Between Clinical, Laboratory and Ultrasonographic Findings With Development of Maternal and Neonatal Complications in Women With Severe Preeclampsia
Brief Title: The Association Between Different Markers With Development of Maternal and Neonatal Complications in Women With Severe Preeclampsia
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Professor, Cairo University
Other Study IDs: 366; Cairo university (Other: Cairo university)
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Severe Preeclampsia
Keywords: preeclampsia; complications
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
pregnant women diagnosed with severe preeclampsia were subjected to • Full history taking including a detailed history of the hypertension state during the current pregnancy (onset, course, current medication, and whether the blood pressure is controlled or not).gravidity , parity mode of delivery any medical disorders, the presence of headache ,blurring of vision and epigastric pain.

* Complete physical examination: general (including BMI & blood pressure measurement) and obstetric examinations.
* Routine obstetric ultrasound and Doppler indices Including umbilical artery Doppler (RI).
* Laboratory investigations :

  1. Complete blood count (CBC). 2 albuminuria will be detected by dipstick kits . 3. Liver enzymes & kidney function. 4.PT,PC,INR.
* Pelvic-Abdominal ultrasound to assess the presence of ascites Ultrasound examination will be performed by a consultant obstetrician to detect free fluid in the peritoneal cavity, especially at hepato-renal pouch, sub-splenic area, or para-colic gutters.

The presence of ascites will be further confirmed at the time of delivery.

3-All labours will be attended by an expert neonatologist and the following will be recorded:

* APGAR score at (1 min).
* The further need for neonatal intensive care unit (NICU) admission.
* Perinatal death

DETAILED DESCRIPTION:
pregnant women diagnosed with severe preeclampsia were subjected to • Full history taking including a detailed history of the hypertension state during the current pregnancy (onset, course, current medication, and whether the blood pressure is controlled or not).gravidity , parity mode of delivery any medical disorders, the presence of headache ,blurring of vision and epigastric pain.

* Complete physical examination: general (including BMI & blood pressure measurement) and obstetric examinations.
* Routine obstetric ultrasound and Doppler indices Including umbilical artery Doppler (RI).
* Laboratory investigations :

  1. Complete blood count (CBC). 2 albuminuria will be detected by dipstick kits . 3. Liver enzymes & kidney function. 4.PT,PC,INR.
* Pelvic-Abdominal ultrasound to assess the presence of ascites Ultrasound examination will be performed by a consultant obstetrician to detect free fluid in the peritoneal cavity, especially at hepato-renal pouch, sub-splenic area, or para-colic gutters.

The presence of ascites will be further confirmed at the time of delivery.

3-All labours will be attended by an expert neonatologist and the following will be recorded:

* APGAR score at (1 min).
* The further need for neonatal intensive care unit (NICU) admission.
* Perinatal death

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age from 18 to 40 years.
2. Gestational age (28_38) weeks, confirmed by the first day of the last menstrual period or first trimesteric ultrasound
3. All suffering of severe preeclampsia

Exclusion Criteria:

1. known liver disease
2. Maternal medical disorders rather than hypertension.
3. Rupture of membrane.
4. Renal disorder.
5. History of illicit drug use.
6. Fetal congenital anomalies.
7. The maternal administration of respiratory depressants within 2 hours from the delivery of the fetus (e. g., opioid analgesic )
8. Associated inflammatory disease or sepsis.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant women with severe preeclampsia
Study Population: All suffering of sever preeclampsia that characterized with one or two of the following:( Dennis A. T etal2012)
  1. Blood pressure of 160/110 or more.
  2. Thrombocytopenia (platelet count less than 100,0000 / microliter).
  3. Impaired liver function (elevated blood levels of liver transaminases to twice the normal concentration).
  4. Severe persistent right upper quadrant or epigastric pain unresponsive to medication and not accounted for by alternative diagnosis, or both.
  5. The new development of renal insufficiency (elevated serum creatinine> 1.1mg/dL or a doubling of serum creatinine in the absence of other renal disease)
Sampling Method: Non-Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Number of participants developed eclampsia | 3 days after delivery
  convulsions in women with severe preeclampsia

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No